CLINICAL TRIAL: NCT05456737
Title: Investigation of Ankle-Foot Characteristics, Balance, Funtional Activity and Quality of Life in Children With Idiopatic Pes Equinovarus
Brief Title: Functional Assessment in Children With Clubfoot
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Özlem Aydın, Physiotherapist, Medipol University
Other Study IDs: 10840098-604.01.01-E.1590 / 56
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Clubfoot
Keywords: Balance; Disability; Foot anthropometry; Pes eqinovarus; Quality of life
MeSH Terms: conditions — Clubfoot | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unilateral Group: Participants with a diagnosis of unilateral clubfoot treated with the Ponseti method were evaluated once with the following evaluation methods:
  Anthropometric measurements FPI-6 Fizyosoft Balance System Functional Activity and Skills Form. OxAFQ-C and OxAFQ-P Kiddy-Kid-Kiddo KINDL
  Interventions: Other: assessment
- Bilateral Group: Participants with a diagnosis of bilateral clubfoot treated with the Ponseti method were evaluated once with the following evaluation methods:
  Anthropometric measurements FPI-6 Fizyosoft Balance System Functional Activity and Skills Form. OxAFQ-C and OxAFQ-P Kiddy-Kid-Kiddo KINDL
  Interventions: Other: assessment
- Healty Group (Control): Healthy participants with normal development were evaluated once with the following evaluation methods:
  Anthropometric measurements FPI-6 Fizyosoft Balance System Functional Activity and Skills Form. OxAFQ-C and OxAFQ-P Kiddy-Kid-Kiddo KINDL
  Interventions: Other: assessment

INTERVENTIONS:
Other: assessment — Application of various assessment methods to determine the foot characteristics, foot posture, functional activity, balance levels and quality of life of the determined groups.

SUMMARY:
The aim of this study was to determine ankle-foot characteristics, load distribution on foot, balance-proprioception, functional activity skills, disability and quality of life levels in children treated with Ponseti's method, finding out the asymetries between both feet in each group, to determine the differences between the healthy foot and the clubfeet, and also to examine the relationship between all parameters in healty children and children with clubfoot.

51 children ages ranging 5 to 15, were included in this study. In order to evaluate foot characteristics, anthropometric measurements were applied. FPI-6 is used for foot posture.Fizyosoft Balance System is used to measure the balance and proprioception. Functional activity were evaluated with Functional Activity and Skills Form. Disability were evaluated with OxAFQ-C and OxAFQ-P and KINDL forms are used to assess quality of life.

DETAILED DESCRIPTION:
Pes Equinovarus (PEV) is one of the complex pediatric foot deformities that has a prevalence of 1-2/1000 live births and requires intensive treatment. The majority of patients with clubfeet have the idiopathic form. Men have a higher risk of exposure with a rate of 2-4/1000 compared to women, and bilateral involvement is present in half of the patients. Each child can be affected at different levels according to their mobility and morphological characteristics. The shape and function of the foot are greatly affected by the four components (CAVE) as adductus in the forefoot, cavus in the midfoot, varus in the hindfoot and equinus deformity in the ankle that make up the complex structure of the disease. It has been reported that children with Pes Equinovarus may experience problems with balance-coordination, gross motor skills and muscle strength due to the complex nature of the disease and an unsuccessful treatment, and also their quality of life may be adversely affected due to difficulties in daily activities.

Treatment of the disease is basically in two ways: operative and/or non-operative (conservative). The main goals of both treatments are to improve the mobility of the foot by correcting the four orthopedic deformities that constitute the complex nature of the disease, and to create a functional, painless, full contact with the ground and not needing modified shoes. The Ponseti method, which is one of the conservative treatment methods that is gold standart for the treatment of clubfoot, is a multi-stage method that requires gentle manipulation, weekly serial casting with a special technique, Achilles tenotomy if necessary, and the use of foot abduction orthosis after casting.

Although the clinical and functional results after Ponseti treatment were promising, deviations in plantar pressure distribution were found as a result of pedobarographic measurements and gait analyzes in unilateral and bilateral feet. It was stated that the dimensions of the unilateral foot were smaller than the contralateral foot, and it was stated that the contralateral foot could have different sizes compared to the normally developing foot. There is no definite judgment about foot anthropometry, due to the existence of studies stating that the sizes of the affected and contra-lateral feet are similar in unilateral involvement.

Balance is another parameter that is stated to be negatively affected depending on foot involvement and the severity of the deformity, but studies examining balance and activity-participation levels are very limited.In addition to studies stating that there is a difference in foot-ankle characteristics, plantar pressure distribution and gross motor skills in children who have received Ponseti treatment, there are also studies stating the opposite. The number of studies on activities of daily living and quality of life is quite limited, and there was any study examining balance and proprioception according to unilateral and bilateral involvement.

For this reason, the aim of this study was to compare the foot-ankle characteristics, plantar pressure distribution, functional activity skills, disability, quality of life and balance-proprioception levels in children treated with the Ponseti method primarily with unilateral-bilateral involvement as well as with children who maintain normal development. To examine the relationship between balance-proprioception involvement and functional activity skills, disability and quality of life in children with clubfoot.

51 children ages ranging 5 to 15, were included in this study. In order to evaluate foot characteristics, anthropometric measurements were applied. FPI-6 is used for foot posture.Fizyosoft Balance System is used to measure the balance and proprioception. Functional activity were evaluated with Functional Activity and Skills Form. Disability were evaluated with OxAFQ-C and OxAFQ-P and KINDL forms are used to assess quality of life.

While performing the statistical analysis of the data and creating the table, the affected foot was defined as the 'inferior' (inf) and the unaffected-contralateral foot as the 'superior' (sup) foot, considering the Dimeglio scores for the superior and inferior foot determination for the unilateral group (UG).

In the bilateral group (BG) and the healthy group (SG), the foot on the side on which they wrote (dominant hand) was called 'superior' and the non-dominant side was called 'inferior', since there was no difference between the Dimeglio scores of the children in both feet.

ELIGIBILITY:
Inclusion Criteria:

1. For the Healty group (control)

   * To be volunteer
   * Being between the ages of 5-15
   * Having signed the informed consent form
   * To be approved by the orthopedist that he does not have any orthopedic problems that would prevent walking, balance and activities of daily living, especially standing
   * Not having any neurological disorders
2. For the Pes Equinovarus groups:

   * To be volunteer
   * Being between the ages of 5-15
   * Having signed the informed consent form
   * To be diagnosed with idiopathic pes equinovarus
   * Being treated primarily with the Ponseti method
   * Being able to stand without support
   * Being able to walk without an assistive device

Exclusion Criteria:

* Having a diagnosis of neurologic clubfoot
* clubfoot associated with severe syndromes such as myelomeningocele or Down syndrome, Larsen, Diastrophic Dysplasia
* Diagnosing congenital joint contractures such as Arthrogryposis Multiplex Congenita
* To have an operative treatment for Pes Echinovarus in the last 1 year
* Refusing to participate in the study

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Clubfoot groups: Diagnosed with idiopathic unilateral and bilateral clubfoot
  Healty group : To be called "healthy" who continue their normal developmental stages and not diagnosed with orthopedic disease.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
OxAFQ-C and OxAFQ-P | January 2020 - February 2021
  The Oxford Ankle-Foot Questionnaire child and parent form (OxAFQ-C and OxAFQ-P) was used to assess disability severity and function associated with foot-ankle problems.
  Response options for each item were rated from never (4), rarely (3), sometimes (2), very often (1) to always (0), indicating how often the problem affected the child.
  Scoring on the 4-field scale is calculated by converting the sum of the field scores to each field's percentage scale (0-100). A higher score for an area represents better function.

SECONDARY OUTCOMES:
Foot lenght | January 2020 - February 2021
  The foot length was determined by taking the footprint on the paper and measuring the distance between the two extreme points on the paper with the help of a tape measure.
Forefoot width | January 2020 - February 2021
  Forefoot width, was determined by taking the footprint on the paper and measuring the distance between first and fifth metatarsal on the paper with the help of a tape measure.
Heel width | January 2020 - February 2021
  Heel width was determined by taking the footprint on the paper and measuring the distance between the two extreme points on heel with the help of a tape measure.
Medial malleol-navicular distance | January 2020 - February 2021
  Medial malleol-navicular distance were measured with the help of a tape measure.
Intermalleolar distance | January 2020 - February 2021
  Intermalleolar distance was determined by measuring the distance between the medial malleolus in both feet with the help of a tape measure in the standing position.
Leg circumference | January 2020 - February 2021
  Leg circumference was determined in a standing position by measuring the circumference of the thickest part of the leg with a tape measure.
FPI-6 | January 2020 - February 2021
  It is a scale that determines foot posture by palpation method. Position of the head of the talus in the hindfoot, inclination under the lateral malleolus, inversion-eversion of the calcaneus; In the forefoot, the talonavicular joint area is evaluated against the medial longitudinal arch structure, and the abduction-adduction of the forefoot is scored between -2 and +2 points.
  * 2,-1 codes for supination of the foot, 0 for neutral, +1,+2 for pronation posture. It was used in this study to evaluate bilateral foot posture.
Fizyosoft Balance System | January 2020 - February 2021
  Fizyosoft Balance System, which was developed by engineers and physiotherapists within the scope of the Tübitak Project, is basically based on the principle of using the Nintendo WiiFit system through a computer by developing software for the purpose of objective balance assessment on the balance board. The developed system evaluates the person's static standing balance, load distributions in each foot, postural sway and proprioception.
  The main issues in the evaluation are the changes in the center of gravity in the x and y axes of the cases with eyes open and closed, the change in postural sway, and the position of the body center of gravity on the feet.In this study, it was used to evaluate static balance, proprioception, and load distribution and transfer in the feet.
Functional Activity and Skills Form | January 2020 - February 2021
  The form, which consists of parameters such as straight walking, toe walking, heel walking, running, squatting, standing on one foot and jumping on one foot, measures the ability of the ankle in functional activities. The scoring system is at the item and subgroup level and no total points are used. For each item, it ranges from 0 (severe reduction / no capacity) to 4 (within normal limits) according to the nature of the movement, and a high score reflects high function.
Kiddy-Kid-Kiddo KINDL | January 2020 - February 2021
  Kiddy-KINDL, Kid-KINDL and Kiddo-KINDL, which is used to evaluate general health-related quality of life in this study, are versions of general health-related quality of life, representing different age groups.
  The Kiddy-KINDL Junior Form is used for young children aged 4-7, the Kid-KINDL Child Form: for children aged 8-12, and the Kiddo-KINDL Adolescent Form is used for children aged 13-16.
  In scoring between 0-100, 0 indicates the worst score, while 100 indicates the best score. A high score is an indicator of good quality of life.
Dimeglio Scoring System | January 2020 - February 2021
  The scale developed by Dimeglio et al. measures the correctability of the foot angularly and determines the severity of the deformity.
  In this study, it was used to determine the severity of the deformity and to determine the superior-inferior foot according to the foot severity.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Aydın, M.Sc., Principal Investigator — Medipol University; Devrim Tarakçı, Assoc. Prof., Study Director — Medipol University
Locations (1):
- Dilbade Special Education and Rehabilitation Center, Istanbul, Eyüp, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu C, Wei J, Yan YB, Shang L, Yang XJ, Huang LY, Lei W. Pedobarographic Analysis following Ponseti Treatment for Unilateral Neglected Congenital Clubfoot. Sci Rep. 2018 Apr 19;8(1):6270. doi: 10.1038/s41598-018-24737-w. PMID 29674653
- [Background] Sangiorgio SN, Ebramzadeh E, Morgan RD, Zionts LE. The Timing and Relevance of Relapsed Deformity in Patients With Idiopathic Clubfoot. J Am Acad Orthop Surg. 2017 Jul;25(7):536-545. doi: 10.5435/JAAOS-D-16-00522. PMID 28574943
- [Background] Gelfer Y, Dunkley M, Jackson D, Armstrong J, Rafter C, Parnell E, Eastwood DM. Evertor muscle activity as a predictor of the mid-term outcome following treatment of the idiopathic and non-idiopathic clubfoot. Bone Joint J. 2014 Sep;96-B(9):1264-8. doi: 10.1302/0301-620X.96B9.33755. PMID 25183601
- [Background] Garcia-Gonzalez NC, Hodgson-Ravina J, Aguirre-Jaime A. Functional physiotherapy method results for the treatment of idiopathic clubfoot. World J Orthop. 2019 Jun 18;10(6):235-246. doi: 10.5312/wjo.v10.i6.235. eCollection 2019 Jun 18. PMID 31259147
- [Background] Cosma D, Vasilescu DE. A Clinical Evaluation of the Pirani and Dimeglio Idiopathic Clubfoot Classifications. J Foot Ankle Surg. 2015 Jul-Aug;54(4):582-5. doi: 10.1053/j.jfas.2014.10.004. Epub 2014 Nov 13. PMID 25458441
- [Result] Dobbs MB, Rudzki JR, Purcell DB, Walton T, Porter KR, Gurnett CA. Factors predictive of outcome after use of the Ponseti method for the treatment of idiopathic clubfeet. J Bone Joint Surg Am. 2004 Jan;86(1):22-7. doi: 10.2106/00004623-200401000-00005. PMID 14711941
- [Result] Zapata KA, Karol LA, Jeans KA, Jo CH. Gross Motor Function at 10 Years of Age in Children With Clubfoot Following the French Physical Therapy Method and the Ponseti Technique. J Pediatr Orthop. 2018 Oct;38(9):e519-e523. doi: 10.1097/BPO.0000000000001218. PMID 29965933
- [Result] Andriesse H, Westbom L, Hagglund G. Motor ability in children treated for idiopathic clubfoot. A controlled pilot study. BMC Pediatr. 2009 Dec 15;9:78. doi: 10.1186/1471-2431-9-78. PMID 20003483
- [Result] Agarwal A, Rastogi A. Anthropometric measurements in Ponseti treated clubfeet. SICOT J. 2018;4:19. doi: 10.1051/sicotj/2018010. Epub 2018 May 25. PMID 29806584
- [Result] Loof E. Additional challenges in children with idiopathic clubfoot: is it just the foot? J Child Orthop. 2019 Jun 1;13(3):245-251. doi: 10.1302/1863-2548.13.190076. PMID 31312263
- See also: journal — http://dergi.totbid.org.tr/uploads/pdf_523.pdf
- See also: journal — https://dergi.totbid.org.tr/abstract.php?lang=tr&id=821